CLINICAL TRIAL: NCT05233254
Title: The Effect of Abdominal Hallowing on Coactivation of Lower Extremity Muscles in Patients With Lumbal Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Asst. Prof., Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-11-2021/23
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Disk Herniated Lumbar; Coordination Lack; Muscle Weakness
Keywords: disc herniation; electromyography; muscle coactivation
MeSH Terms: conditions — Ataxia; Muscle Weakness; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with L4-5 disc herniation (Experimental): In the light of the reference research, it was estimated that it could reach an effect size of 0.6 according to the sample size measurement made with at least 80% power and 0.05 margin of error, and 18 individuals with LDH (9 men, 9 women) were planned to participate in this study. Since data loss was predicted to be 20%, it was decided to include a total of 22 patients for the study.
  Interventions: Behavioral: Abdominal Hollowing exercise

INTERVENTIONS:
Behavioral: Abdominal Hollowing exercise — Gently and slowly draw in your lower abdomen below your navel without moving your upper stomach, back and pelvis. Breathe in and out. Gently and slowly draw in your lower abdomen below your navel without moving your upper stomach, back and pelvis. Breathe in and out.

SUMMARY:
Intervertebral disc degenerations are the most important cause of chronic low back pain resulting in job loss and associated socio-economic problems in developed and developing industrial countries 1. More than 40% of the Turkish population has experienced low back pain at least once in their life 2. Intervertebral disc degenerations Lumbal Disc Herniation (LDH), which is frequently represented, can cause motor and sensory losses in the lower extremity by compressing the spinal nerves. Lumbar disc surgery procedure is inevitable in case of advanced functional losses in the related sensory dermatomes and muscles after LDH. Lumbal disc surgeries are performed for the purpose of decompression of nerve pressures on nerves due to advanced disc herniation. they suggest 4.

One of the most common LDH problems in the community is low foot problems due to weakness of the tibialis anterior muscle, which occurs due to L4-L5 disc herniation, and the accompanying functional disorders. In disc herniations at this level, the activation of the tibialis anterior muscle, which is compressed by the nerve root, decreases compared to the medial gastrocnemius muscle, where it works as an antagonist, and this leads to functional limitations, especially in gait and balance activities.

Spinal stabilization exercises are a concept that emerged from the idea that exercise is important for the provision and preservation of functionality of people with low back and back pain due to LDH. According to this exercise approach, muscles are of great importance in providing lumbar region stability. These muscles are classified as general (global) stabilizing muscles, which are dynamic, phasic, and power-producing muscles, and regional (local) stabilizing muscles, which are postural, tonic, and stabilizer muscles. The main muscles responsible for spine stabilization are multifidus, transversus abdominus and pelvic floor muscles 6. It is argued that increased lumbo-pelvic motor control thanks to spine stabilization facilitates lower extremity activities, especially flexion and extension movements in the sagittal plane. Patients with LDH who increase their motor strength can use lower extremity movements more functionally.

The aim of this study was to (1) determine the activation rates of the tibialis anterior and medial gastrocnemius muscles during different functional activities in the lower extremities affected and unaffected by LDH, (2) to compare the rates of the affected extremity to the rates of the healthy extremity during coactivation of the transversus abdominus and multifidus muscles (spinal stabilization basic exercise). to determine whether it is close or not. According to the hypothesis of this study, the researchers thought that the functional activities performed together with the activation of the transversus abdominus and multifidus muscles would show coactivation behaviors at a rate closer to the healthy extremity.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* To be diagnosed with LDH at the minimum level of protrusion by the physician
* Diagnosis confirmed by the physician in charge of the study by computed tomography (CT) or magnetic resonance imaging (MRI) reports

Exclusion Criteria:

* Having bilateral LDH findings,
* have an acute illness
* Having significant neurological disease other than LDH (such as head trauma, brain abscess, brain tumor, migraine attack, seizure)
* Having trauma or congenital orthopedic disorders that prevent lower extremity functions other than LDH
* Not being able to adapt to the study cognitively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Electromyography | 15 minutes
  The non-invasive superficial EMG system (Noraxon USA, Inc., Scottsdale, AZ) will be used to measure activation levels of the tibialis anterior and medial gastrocnemius muscles. Bipolar Ag/AgCl surface electrodes will be placed at intervals of 1 cm and 2 mm between the electrodes. The bandwidth of the processed EMG signals is 20-450 Hz. and input impedances will be limited to greater than 10 mV. The processing rate of EMG data is 1000 Hz. It will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Üniversitesi, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No